CLINICAL TRIAL: NCT04843267
Title: A Multi-center, Non-randomized, Open-label Phase II Clinical Study on the Treatment of Newly Diagnosed Advanced Hodgkin's Lymphoma With PD-1 Antibody (Tislelizumab) Combined With AVD Regimen (Doxorubicin, Vindesine, Dacarbazine) Under the Guidance of PET/CT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-324-01
Record Dates: First submitted 2021-04-12; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Hodgkin Lymphoma; Chemotherapy Effect
MeSH Terms: conditions — Hodgkin Disease | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab in first-line treatment of Hodgkin's lymphoma

SUMMARY:
The experimental drug regimen in this study includes a PD-1 antibody (tislelizumab) single-drug induction treatment period and a PD-1 antibody + AVD combined treatment period.

1. PD-1 antibody (tislelizumab) single-drug induction treatment period (first 2 courses for all patients + 3-6 courses for CR patients):

   PD-1 antibody (tislelizumab), specification: 100mg/bottle. Usage and dosage: intravenous drip, 200mg each time, QD, D1. In the above PD-1 antibody single-drug regimen, 21 days are regarded as a treatment cycle, and all patients first receive 2 courses of PD-1 antibody single-drug induction treatment;
2. PET/CT mid-term efficacy evaluation used for guiding follow-up treatment options:

   PET/CT efficacy evaluation before the 3rd course of treatment (PET/CT2):

   CR patients: continue to receive PD-1 antibody monotherapy, and then receive 4 courses of PD-1 antibody therapy; PR patients: sequential 4 courses of PD-1 antibody + AVD combined chemotherapy; PD+SD patients: out group, and receive other anti-lymphoma therapy deemed suitable by the investigators;

   After the 6th course, patients not out of the group receive PET/CT3 efficacy evaluation:

   CR patients: end the treatment and enter the follow-up; PR patients: receive 2 more courses of PD-1 antibody + AVD combined chemotherapy, and then enter the follow-up.
3. PD-1 antibody + AVD combined treatment period (3rd-6th/8th course for PR patients):

PD-1 antibody, specification: 100mg/bottle. Usage and dosage: intravenous drip, 100mg each time, QD, d1, d15. AVD regimen Doxorubicin 25mg/m2, d1, d15 intravenous injection Vindesine 3mg/m2, d1, d15 intravenous injection Dacarbazine 0.375mg/m2, d1, d15 intravenous drip In this combined treatment regimen, every 28 days is a treatment cycle, and the PD-1 antibody is used in combination with AVD in D1 and D15 of each treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed classical Hodgkin lymphoma (HL) confirmed by histopathology;
2. Stage III-IV, or Stage IIB patients with at least one high-risk factor (NCCN standard)
3. Patients not suitable for receiving radiotherapy subsequently
4. Patients with at least one assessable lesion (according to Lugano 2014 standard);
5. Age 18 or above (including 18), no gender requirement;
6. ECOG PS score of 0-1 points;
7. Expected survival time ≥ 3 months;
8. Hematopoietic function: absolute neutrophil count ≥ 1.5×109/L, platelets ≥ 90×109/L, hemoglobin ≥ 90g/L; liver function: for patients with non-hepatitis B, total bilirubin, ALT and AST <1.5×ULN (upper limit of normal); patients with hepatitis B need to take effective antiviral drugs, and HBV-DNA copy <2000 IU/ml and ALT<2×ULN; renal function: creatinine <1.5×ULN and creatinine clearance rate ≥50ml/min;
9. With normal main indicators of cardio-pulmonary function, and no obvious contraindication to chemotherapy;
10. Not received any anti-tumor therapy such as radiotherapy, chemotherapy, targeted therapy, cellular immunotherapy or hematopoietic stem cell transplantation before enrollment;
11. Voluntarily signing an informed consent form before trial screening.

Exclusion Criteria:

1. Nodular lymphocyte predominant HL;
2. Patients received any form of anti-tumor therapy in the past;
3. Patients planning to receive radiotherapy or autologous stem cell transplantation;
4. With involvement of central nervous system (meninges or brain parenchyma);
5. Pregnant and lactating women and child-bearing patients who are unwilling to take contraceptive measures;
6. Patients with history of other tumors, except for cured cervical cancer orskin basal cell carcinoma; patients who have received organ transplantation;
7. Patients who have received symptomatic treatment of myelosuppressive toxicity within 7 days before enrollment;
8. Patients who have used any immunosuppressive drugs within 4 weeks before the first-dose treatment,
9. Patients with known active interstitial pneumonia;
10. Abnormal liver function (total bilirubin>1.5×ULN, ALT/AST>2.5×ULN or ALT/AST>5×ULN for patients with liver invasion), abnormal renal function (serum creatinine>1.5×ULN), abnormal electrolyte metabolism;
11. Peripheral neuropathy ≥ Grade 2;
12. Patients with a history of prolonged QT interval which is of clinical significance (male> 450ms, female> 470ms), ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI) within 1 year, congestive heart failure (CHF), patients with symptomatic coronary heart disease requiring drug therapy;
13. Patients with the end-diastolic width of fluid sonolucent area in pericardial cavity ≥10mm by cardiac B-ultrasonography;
14. Mentally disturbed/patients unable to give informed consent;
15. Patients who affect the evaluation of test results due to drug abuse or long-term alcohol abuse;
16. Participating in another interventional clinical study at the same time; Patients not suitable to participate in this trial by the judgment of investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
complete response rate after two cycles of tislelizumab | 6 weeks
  complete response rate after two cycles of tislelizumab by PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No